CLINICAL TRIAL: NCT03829436
Title: A Phase 1/1b Open-label, Dose-escalation and Dose-expansion Study of TPST-1120 as a Single Agent or in Combination With Systemic Anti-Cancer Therapies in Subjects With Advanced Solid Tumors
Brief Title: TPST-1120 as Monotherapy and in Combination With Nivolumab in Subjects With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tempest Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TPST-1120-001
Record Dates: First submitted 2019-01-30; First posted 2019-02-04 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma; Metastatic Castration Resistant Prostate Cancer; Renal Cell Carcinoma; Non-small Cell Lung Cancer; Colorectal Cancer; Squamous Cell Carcinoma of Head and Neck; Triple-Negative Breast Cancer; Urothelial Carcinoma; Cholangiocarcinoma; GastroEsophageal Cancer; Pancreatic Cancer; Sarcoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Cholangiocarcinoma; Pancreatic Neoplasms; Sarcoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 TPST-1120 (Experimental): Subjects will receive escalating doses of TPST-1120 administered orally twice daily continuously until MTD is reached or until disease progression
  Interventions: Drug: Part 1 TPST-1120
- Part 2 TPST-1120 + nivolumab (Experimental): Subjects will receive escalating doses of TPST-1120 administered orally twice daily in combination with nivolumab administered intravenously every 28 days until MTD is reached for TPST-1120 or until disease progression.
  Interventions: Drug: Part 2 TPST-1120 + nivolumab
- Part 3 TPST-1120 (Experimental): Selected dose of TPST-1120 administered orally twice daily until disease progression
  Interventions: Drug: Part 3 TPST-1120
- Part 4 TPST-1120 + nivolumab (Experimental): Selected dose of TPST-1120 administered orally twice daily in combination with nivolumab administered intravenously every 28 days until MTD is reached for TPST-1120 or until disease progression
  Interventions: Drug: Part 4 TPST-1120 + nivolumab

INTERVENTIONS:
Drug: Part 1 TPST-1120 — Subjects will receive escalating doses of TPST-1120 administered orally twice daily continuously until MTD is reached or until disease progression
  Other Names: Experimental
  Arms: Part 1 TPST-1120
Drug: Part 2 TPST-1120 + nivolumab — Subjects will receive escalating doses of TPST-1120 administered orally twice daily
  Other Names: Experimental + Opdivo
  Arms: Part 2 TPST-1120 + nivolumab
Drug: Part 3 TPST-1120 — Selected dose of TPST-1120 administered orally twice daily until disease progression
  Other Names: Experimental
  Arms: Part 3 TPST-1120
Drug: Part 4 TPST-1120 + nivolumab — Selected dose of TPST-1120 administered orally twice daily in combination with nivolumab administered intravenously every 28 days until MTD is reached for TPST-1120 or until disease progression
  Other Names: Experimental + Opdivo
  Arms: Part 4 TPST-1120 + nivolumab

SUMMARY:
This is a phase 1/1b open label, multicenter dose escalation and dose expansion study to investigate the safety, tolerability and anti-tumor activity of TPST-1120, a small molecule selective antagonist of PPARα (peroxisome proliferator activated receptor alpha) as monotherapy and in combination with a systemic anticancer agent, nivolumab, an anti-PD1 antibody, in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a phase 1/1b open label, multicenter, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of TPST-1120, a small molecule selective antagonist of PPARα (peroxisome proliferator activated receptor alpha) in adult subjects with selected advanced solid tumors. TPST-1120 will be administered as monotherapy and in combination with a systemic anticancer agent, nivolumab, an anti-PD1 antibody, in subjects with advanced solid tumors. This trial is composed of dose escalation and dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria

* Eastern Cooperative Oncology Group performance status of 0-1 at enrollment
* Progressive disease or previously untreated tumors for which no standard therapy exists or treatment naïve at the time of study entry are eligible
* Have at least one measurable lesion according to RECIST v1.1
* Subjects with the following histologies are eligible and who are refractory to, have failed, are intolerant to, are ineligible for standard therapy, or for which no standard therapy exists are eligible: Part 1 (Dose Escalation- Monotherapy): RCC, NSCLC, CRC, metastatic castration resistant prostate cancer (mCRPC), cholangiocarcinoma, TNBC, pancreatic cancer, HCC, gastroesophageal cancer, squamous cell carcinoma of head and neck (SCCHN), urothelial bladder cancer (UBC), and sarcoma (liposarcomas and leiomyosarcomas); Part 2 (Dose Escalation-Combination with nivolumab): RCC, HCC, and cholangiocarcinoma; Part 3 (Dose Expansion-Monotherapy): RCC, HCC and cholangiocarcinoma; Part 4 (Dose Expansion-Combination with nivolumab): HCC.

Exclusion Criteria

* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study, a specimen-collection study or the follow-up period of an interventional study
* Any chemotherapy, monoclonal antibody therapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment within 28 days of commencing TPST-1120 treatment. Targeted therapy such as tyrosine kinase inhibitors within 14 days of commencing first dose of study drug(s)
* For subjects who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA4 therapy:

  1. Subjects must not have experienced an irAE toxicity that led to permanent discontinuation of prior immunotherapy.
  2. Any unresolved irAE > Grade 1 with prior immunotherapy treatment.
* Symptomatic, untreated or actively progressing central nervous system metastases
* Have received fibrates within 28 days before first dose of investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) of TPST-1120 as a single agent and in combination with nivolumab. | From start of treatment to end of treatment, up to 36 months
  Incidence of dose limiting toxicities (DLTs) of TPST-1120 as a single agent and in combination with nivolumab.
Incidence of treatment-emergent adverse events as assessed by NCI-CTCAE v5.0 of TPST-1120 as a single agent and in combination with nivolumab. | From start of treatment to end of treatment, up to 36 months
  Incidence of treatment-emergent adverse events as assessed by NCI-CTCAE v5.0 of TPST-1120 as a single agent and in combination with nivolumab.
Identify the maximum tolerated dose | From start of treatment to end of treatment, up to 36 months
  Incidence of dose limiting toxicities (DLTs) of TPST-1120 as a single agent and in combination with nivolumab.

SECONDARY OUTCOMES:
Assess pharmacokinetics: Maximum serum concentration (Cmax) | Day 1, 2, 8 of Cycle 1 and Day 1 of Cycle 3 (cycle can be 21 or 28 days, depending on cohort assignment)
  Maximum serum concentration (Cmax) of TPST-1120
Assess pharmacokinetics: Area under the curve (AUC) | Day 1, 2, 8 of Cycle 1 and Day 1 of Cycle 3, Day 1 of Cycles 5+ (cycle can be 21 or 28 days, depending on cohort assignment)
  Area under the curve (AUC) of TPST-1120
Objective response rate | From start of treatment to end of treatment, up to 36 months
  Objective response rate per RECIST v1.1 criterion of TPST-1120 as a single agent and in combination with nivolumab.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stagg, PharmD, Study Director — Tempest Therapeutics
Locations (11):
- United States (11):
  - University of California - San Francisco, San Francisco, California
  - Miami Cancer Institute, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute - TN, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No